CLINICAL TRIAL: NCT07239414
Title: Bempedoic Acid Versus Statins in Primary-Prevention Patients With Suboptimal Statin Adherence: Effects on LDL-C Reduction and Tolerability
Acronym: BASIS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sohaib Ashraf (Other)
Responsible Party: Sponsor-Investigator, Sohaib Ashraf, Consultant Cardiologist, Sheikh Zayed Federal Postgraduate Medical Institute
Organization: Sheikh Zayed Federal Postgraduate Medical Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RAIC PESSI/ESTT/2025/506
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular
Keywords: bempodoic acid
MeSH Terms: interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Tablets; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Bempedoic acid) (Active Comparator): BA 180 mg once daily + placebo statin.
  Interventions: Drug: Bempedoic Acid 180 MG Oral Tablet; Drug: Placebo
- Arm B (Statin) (Placebo Comparator): Rosuvastatin 5 mg once daily + placebo BA.
  Interventions: Drug: Rosuvastatin 5 mg; Drug: Placebo

INTERVENTIONS:
Drug: Bempedoic Acid 180 MG Oral Tablet — BA 180mg OD
  Arms: Arm A (Bempedoic acid)
Drug: Rosuvastatin 5 mg — rosuvastatin 5mg HS
  Arms: Arm B (Statin)
Drug: Placebo — Placebo given OD

SUMMARY:
Bempedoic acid is an oral, non-statin LDL-cholesterol (LDL-C) lowering agent that inhibits ATP citrate lyase (ACL), upstream of HMG-CoA reductase (the enzyme inhibited by statins).

MDPI

+1

In patients with hypercholesterolemia who are unable to tolerate statins, or have sub-optimal statin adherence/tolerance, bempedoic acid has been shown to reduce LDL-C by ~20-30% (monotherapy) and more when added to other therapies (e.g., ezetimibe) (≈30-40%).

PubMed

* 2 medicinejournal.in
* 2

In the large primary-prevention subgroup of the trial CLEAR Outcomes (statin-intolerant patients without prior cardiovascular event), bempedoic acid (180 mg daily) lowered LDL-C by ~21.3% and hs-CRP by ~21.5%. It also was associated with a significant reduction in major adverse cardiovascular events (MACE): hazard ratio 0.70 (95% CI 0.55-0.89) versus placebo over ~40 months.

PubMed +1

Regarding tolerability: muscle-related adverse events appear lower compared to statins (because bempedoic acid is activated only in the liver, not in skeletal muscle) and it appears generally well tolerated, but there are signals of increased uric acid/gout, elevated hepatic enzymes, and creatinine/renal effects.

MDPI

+1

Comparative cardiovascular benefit (when normalized per unit LDL-C reduction) suggests that bempedoic acid may yield similar relative risk reductions as statins, though absolute LDL-C lowering is less.

DETAILED DESCRIPTION:
Mechanism: Bempedoic acid works by inhibiting ACL in the cholesterol-synthesis pathway; since the activating enzyme is present only in the liver (not muscle), the risk of muscle-related side-effects is diminished.

Frontiers

Indication/Use Case: Particularly useful in patients who (a) are at elevated cardiovascular risk (primary prevention or secondary), (b) cannot tolerate statins or have suboptimal adherence, and (c) need further LDL-C reduction beyond statin (or in place of statin) therapy.

Efficacy:

~20-30% LDL-C lowering as monotherapy in statin-intolerant patients. PubMed

+1

Additional benefit when combined with other therapies (e.g., ~30-40% reduction when combined with ezetimibe).

medicinejournal.in

In primary-prevention high-risk patients intolerant of statins: LDL-C reduction ~21% and hs-CRP ~21% with meaningful reduction in cardiovascular events.

PubMed +1

Tolerability/Safety:

Lower risk of muscle symptoms compared to statins. PubMed

+1

Known adverse signals: hyperuricemia/gout, elevated liver enzymes, possibly increased creatinine/renal changes.

JAMA Network +1

Comparison with Statins:

Statins typically reduce LDL-C by much larger margins (30-50%+ depending on dose/intensity). Bempedoic acid's LDL-C reduction is more modest in comparison.

However, when looking at the risk reduction per unit LDL-C lowering, bempedoic acid appears to yield similar relative benefits as statins.

American College of Cardiology

+1

Clinical Implication: In patients with suboptimal statin use (due to intolerance, non-adherence, or contraindication), bempedoic acid offers a viable adjunct or alternative lipid-lowering strategy in the primary prevention setting.

Limitations:

Not a direct head-to-head trial of bempedoic acid versus statins in the scenario of suboptimal statin adherence.

Absolute reduction in LDL-C is lower than high-intensity statins, so expectations must be calibrated accordingly.

Long-term safety in wider populations continues to be monitored.

Cost and accessibility may vary by region; local cost-effectiveness needs evaluation.

ELIGIBILITY:
Inclusion Criteria

* Adults aged ≥40 years with no established ASCVD (no prior myocardial infarction, stroke, or acute coronary syndrome).
* Indicated for lipid-lowering therapy (LDL-C ≥130 mg/dL or 10-year ASCVD risk

  ≥7.5%).
* Documented history of poor statin adherence, defined as:

  * Self-reported adherence <80% in the past 3 months, or
  * Prior statin discontinuation for adverse effects documented in the medical record.
* Willingness to provide written informed consent. Exclusion Criteria
* Established ASCVD (secondary prevention).
* Severe hepatic impairment (ALT or AST >3× upper limit of normal).
* Severe renal impairment (eGFR <30 mL/min/1.73 m²).
* Pregnancy, breastfeeding, or women of childbearing potential not using contraception.
* Current or planned treatment with PCSK9 inhibitors, fibrates, or niacin.
* Known hypersensitivity to study drugs or excipients.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Estimated)
Dates: Start 2025-11-10 (Estimated); Primary Completion 2026-11-10 (Estimated); Study Completion 2027-02-21 (Estimated)

PRIMARY OUTCOMES:
Percentage change in LDL-C | 6 months
  Percentage change in LDL-C from baseline LDL-C
Composite adherence/tolerability endpoint: | 6 months
  treatment discontinuation, muscle-related symptoms, or laboratory abnormalities (ALT/AST >3× ULN, uric acid >9 mg/dL).

SECONDARY OUTCOMES:
Absolute change in LDL-C | 6 months
  Absolute change in LDL-C from baseline to 6 months.
Proportion achieving LDL-C <100 mg/dL (or <70 mg/dL for diabetics). | 6 months
  Proportion achieving LDL-C <100 mg/dL (or <70 mg/dL for diabetics).
Change in hs-CRP | 6 months
  Change in hs-CRP from baseline.

IPD SHARING:
Plan to Share IPD: Undecided